CLINICAL TRIAL: NCT00916201
Title: Evaluation of Potential Central Glucoregulatory Compounds to Treat/Ameliorate the Symptoms of Schizophrenia: a Proof-of-concept Study in Healthy Volunteers.
Brief Title: Evaluation Study of New Compounds With Potential Use in Schizophrenia
Acronym: EICAS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Max Planck Institute for Metabolism Research (Other)
Responsible Party: Principal Investigator, F Markus Leweke, Professor, Central Institute of Mental Health, Mannheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EICAS
Record Dates: First submitted 2009-05-05; First posted 2009-06-09 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — cyclohexyl carbamic acid 3'-carbamoylbiphenyl-3-yl ester

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intranasal Insulin (Experimental): Intranasal administered insulin
  Interventions: Drug: intranasal Insulin
- Cannabidiol CR (Experimental): Cannabidiol is the main non psychoactive compound of the Cannabis sativa plant.
  Interventions: Drug: Cannabidiol CR
- URB597 (Experimental): URB597 is a selective inhibitor of the Fatty acid amide hydrolase enzyme.
  Interventions: Drug: URB597

INTERVENTIONS:
Drug: URB597 — 10 mg / d for 5 days, orally
  Arms: URB597
Drug: intranasal Insulin — 160 IU / d for 5 days, intranasal
  Arms: Intranasal Insulin
Drug: Cannabidiol CR — 320 mg / d for 5 days, orally
  Other Names: Arvisol
  Arms: Cannabidiol CR

SUMMARY:
Different compounds that might modify the glucose regulation in the central nervous system will be evaluated in healthy volunteers. Several examinations will be performed in order to get a detailed plan how these substances might work.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Informed consent given by the subject
* Both, female and male subjects may participate
* Age between 18 and 65 years
* Negative drug-screening at the time of screening
* In female participants in fertile age, reliable contraception, which means contraception's pearl-index is equal or smaller than 1.
* Non-Smoker
* Body Mass Index between 18 and 40.

Exclusion Criteria:

* Lack of accountability
* Any current psychiatric disorder through the Structured Clinical Interview for DSM-IV (SCID) at the time of screening
* Any known psychiatric or neurological illness in the participant's history.
* Known family history concerning psychiatric disorders
* Relevant use of cannabis (which is defined on the present state of knowledge as at the most five times lifetime-consumption and no consumption for at least one year)
* Pregnancy or lactation phase in female at the time of screening
* Severe physical (internal) or neurological illness, especially cardiovascular, renal, advanced respiratory, haematological or endocrinological failures or infectious diseases (acute hepatitis A, B or C or HIV) assessed at the time of the screening by the subject's history, clinical examination and laboratory testing, at the discretion of the investigator
* Consumption of any illegal drugs (except cannabis in history, see above)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Clinical assessment with several psychopathological scores for self-assessment and peer evaluation (BPRS, PANSS, SIPS, CGI, MADRS, HAM-A, SCL-90-R) | Seven days
Laboratory assessment (routine testing, "-omics", genetic analyses, endocannabinoid levels) | Seven days
Diagnostics of the cerebrospinal fluid | Seven days
fMRI scan of the brain | Seven days

SECONDARY OUTCOMES:
Regular evaluating of the subject's condition and ability to continue the study by CGI | Seven days
Regular laboratory testing and ECG | Seven days
Scales for the assessment of adverse events (UKU, SCL- 90-R) | Seven days
(Numbers of) SAE and AE | Seven days

CONTACTS AND LOCATIONS:
Overall Officials: F. Markus Leweke, MD, Principal Investigator — Central Institute of Mental Health
Locations (1):
- Dep. of Psychiatry and Psychotherapy, Central Institute of Mental Health, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No